CLINICAL TRIAL: NCT02819102
Title: A Single Sequence, Open-Label Drug-Drug Interaction Study to Evaluate the Effect of BCX7353 on Cytochrome P450 3A4, 2C9, 2C19 and 2D6 Enzyme Activity Using Probe Substrates in Healthy Subjects
Brief Title: An Open-label Drug-Drug Interaction Study to Evaluate the Effect of BCX7353 on Cytochrome P450 Enzyme Activity Using Probe Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX7353-102
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-06

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metabolic Probes and BCX7353 (Experimental): Day 1: 1 mg midazolam will be administered as an IV bolus simultaneously to administration of 500 mg tolbutamide, 40 mg omeprazole, and 30 mg dextromethorphan orally.
  Day 2: a single oral dose of 2 mg midazolam. Days 3 to 9: 350 mg BCX7353 once a day. Day 10: 1 mg midazolam will be administered as an IV bolus simultaneously to administration of 500 mg tolbutamide, 40 mg omeprazole, 30 mg dextromethorphan and 350 mg BCX7353, orally.
  Day 11: a single oral dose of 2 mg of midazolam along with 350 mg BCX7353.
  Interventions: Drug: BCX7353 and probes

INTERVENTIONS:
Drug: BCX7353 and probes

SUMMARY:
This is an open-label, single sequence study to evaluate the effect of BCX7353 on hepatic and intestinal cytochrome P450 enzymes using probe substrate drugs in healthy subjects. Pharmacokinetics of the probe substrate drugs will be measured prior to and following administration of multiple doses of BCX7353.

DETAILED DESCRIPTION:
This is a single centre, single sequence, open-label, study to evaluate the effect of BCX7353 on hepatic and intestinal cytochrome P450 (CYP) 3A4 (midazolam IV and PO, respectively), CYP2C9 (tolbutamide), CYP2C19 (omeprazole) and CYP2D6 (dextromethorphan) enzyme activity using probe substrate drugs in healthy subjects. Pharmacokinetics of the probe substrate drugs will be measured prior to and following administration of multiple doses of BCX7353.

Twenty healthy male and female subjects are planned for dosing.

Each subject will receive the following treatments:

Day 1: 1 mg midazolam will be administered as an IV bolus simultaneously to administration of 500 mg tolbutamide, 40 mg omeprazole, and 30 mg dextromethorphan orally.

Day 2: a single oral dose of 2 mg midazolam. Days 3 to 9: 350 mg BCX7353 once a day. Day 10: 1 mg midazolam will be administered as an IV bolus simultaneously to administration of 500 mg tolbutamide, 40 mg omeprazole, 30 mg dextromethorphan and 350 mg BCX7353, orally.

Day 11: a single oral dose of 2 mg of midazolam along with 350 mg BCX7353.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Body mass index 18 to 32 kg/m2
* Abides by study restrictions
* Attends all study visits and agrees to remain in study center for the confinement period
* Acceptable birth control measures for male subjects and women of childbearing potential

Key Exclusion Criteria:

* Clinically significant medical history, current medical or psychiatric condition. This includes a history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, or cardiac disease
* Clinically significant ECG finding, vital sign measurement or laboratory/urinalysis abnormality at screening or baseline
* Poor or ultra- metabolizers of CYP2C19 or CYP2D6 Use of over the counter or prescription medication within 14 days of dosing and anticipated use through the follow-up visit
* Use of medication or consumption of any substance that is known to inhibit or induce metabolic enzymes or transporters within 30 days of dosing
* Participation in any other investigational drug study within 90 days of screening
* Recent or current history of alcohol or drug abuse
* Regular recent use of tobacco or nicotine products
* Positive serology for HBV, HCV, or HIV
* Pregnant or nursing
* Donation or loss of greater than 400 mL of blood within 3 months
* Serious adverse reaction or serious hypersensitivity to any drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cmax of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
Tmax of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
AUClast of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
AUCinf of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
t1/2 of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
Cl of intravenous midazolam | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11

SECONDARY OUTCOMES:
adverse events | absolute and change from baseline through study day 11
laboratory analyses | absolute and change from baseline through study day 11
Vital signs | absolute and change from baseline through study day 11
physical examination findings | absolute and change from baseline through study day 11
electrocardiograms | absolute and change from baseline through study day 11
C24 for tolbutamide | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
C6 for IV and oral midazolam | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
Probe/metabolite AUC24 ratio | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
Tlag of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
VdF of probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
CL/F of oral probe substrates | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11
Vss of intravenous midazolam | plasma pharmacokinetic parameters are based on blood sampling through 24 hours on Day 1, 2, 10 and 11

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Ruddington, Nottingham, United Kingdom